CLINICAL TRIAL: NCT01504490
Title: A Phase I Study of a Combination of the Proteosome Proliferator-Activated Receptor Gamma Agonist, CS-7017 and the Retinoid X Receptor Agonist, Bexarotene
Brief Title: Phase I Study of CS-7017 and Bexarotene
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug no longer available
Sponsor: Georgetown University (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-345
Record Dates: First submitted 2011-12-14; First posted 2012-01-05 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Solid Tumors; Lymphoma; Multiple Myeloma
Keywords: Advanced cancer
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — efatutazone; Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CS-7017 and Bexarotene (Experimental): Combination of CS-7017 and Bexarotene
  Interventions: Drug: CS-7017 and Bexarotene

INTERVENTIONS:
Drug: CS-7017 and Bexarotene — CS-7017 will be administered orally, twice daily for 28 days of each 28-day cycle in escalating doses depending on cohort patient is assigned to.
  Bexarotene will be administered orally once daily for 28 days of each 28-day cycle. The dose a patient receives will depend on which cohort the patient is assigned to.
  Other Names: Efatutazone; Targretin

SUMMARY:
This study is for patients with advanced solid tumors. The purpose of this study is to test the safety and effectiveness of a new combination of drugs, CS-7017 and Bexarotene in patients with advanced cancer. CS-7017 and Bexarotene both have many effects on cancer cells, including stopping cancer cells from growing and dividing, and causing the cancer cells to die. CS-7017 and Bexarotene work on cancer cells in a similar manner and both drugs together may have an even greater effect against cancer cells, hopefully, increasing the killing of cancer cells.

CS-7017 is an investigational or experimental anti-cancer agent that has not yet been approved by the Food and Drug Administration (FDA) for use in any type of cancer. Bexarotene is an anti-cancer agent that has been approved by the FDA for patients with a specific type of cancer, cutaneous T-cell lymphoma.

This study will help find out what effects the combination of drugs, CS-7017 and Bexarotene, has on cancer. This research is being done because it is not known if CS-7017 is safe to be given with Bexarotene.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced malignancy with measurable disease except for acute leukemias
* Progression on, or intolerance of, or ineligibility for all standard therapies
* Biopsy accessible tumor deposits
* LVEF >/= institutional normal
* No evidence of clinically significant fluid retention
* ECOG Performance status 0-2
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated with surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of intracranial disease and have not had treatment with steroids within one week of study enrollment.
* Adequate hepatic, bone marrow, and renal function
* Partial thromboplastin time must be </= 1.5 x upper limit of normal range and INR < 1.5. Subjects on anticoagulant will be permitted to enroll as long as the INR is in the acceptable therapeutic range
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Subject is capable of understanding and complying with parameters of the protocol and able to sign and date the informed consent.

Exclusion Criteria:

* Prior CS-7017 treatment
* Treatment with thiazolidinediones (TZDs) within 4 weeks prior to start of study treatment
* Current need for concomitant use of other TZDs during the study
* Grade 2 or greater fasting hypertriglyceridemia
* Concurrent use of insulin
* Concurrent use of known CYP 3A4 inhibiting or activating medications
* CNS metastases which do not meet the criteria outlines in inclusion criteria
* Active severe infection or known chronic infection with HIV or hepatitis B virus
* Cardiovascular disease including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke or congestive heart failure within the last 6 months
* Life-threatening visceral disease or other severe concurrent disease
* Women who are pregnant or breastfeeding
* Anticipated survival under 3 months
* Clinically significant and uncontrolled major medical condition(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  The highest dose at which < 1 out of 6 subjects experienced a dose-limiting toxicity

SECONDARY OUTCOMES:
Response rate | 4 months
  Complete response + partial response
Disease control rate | 4 months
  Response rate + stable disease
Pharmacodynamic effects | Prior to treatment, Just prior to Day 1 and just prior to Day 15 of cycle 1
  PPAR-gamma and RXR analysis by immunohistochemistry; Tumor staining for the following PPAR-gamma regulated genes: Cyclin D1, p16, p18, p21, p27, and c-myc.
Pharmacokinetics | Day -7 prior to first dose of CS-7017, Day 1, and Day 15 of Cycle 1
  Trough serum levels of CS-7017 and its metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States